CLINICAL TRIAL: NCT03351907
Title: Prospective Cohort Study of Cardiovascular Disease in Guangdong Province
Brief Title: Cardiovascular Disease Cohort in Guangdong Province
Status: Active, not recruiting | Type: Observational
Sponsor: Min Xia (Other)
Responsible Party: Sponsor-Investigator, Min Xia, Professer, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 2017XXG1120
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Urine and fecal samples for biochemical tests, biomarker examination and DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with cardiovascular diseases from Guangdong province will be recruited and followed up for at least 4 years to evaluate the risk factors for cardiovascular-related mortality and disability. Physical examination, questionnaire survey and biological sample collection will be conducted at baseline and the incidence of all-cause and cardiovascular mortality will be investigated during follow-up.

DETAILED DESCRIPTION:
5,000 patients (30-85 years old) with primary hypertension, coronary heart disease, heart failure or peripheral vascular disease and who have been living in Guangdong province for more than 5 years will be recruited. All participants will be prospectively followed up for the incidence of all-cause and cardiovascular mortality. Information about socio-demographic, diet, lifestyle, psychological status, medical history and current medication will be collected by questionnaires. Physical examinations including height, weight, waist and hip circumferences, blood pressure, fat mass and vital capacity will be conducted.Besides, blood, urine and fecal samples will be collected for further analysis. The associations between diet and lifestyle and risks for cardiovascular disease will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular disease patients (30-85 years old) who have been living in Guangdong province for more than 5 years.
* Patients have been diagnosed with primary hypertension, coronary heart disease, heart failure or peripheral vascular disease, etc.

Exclusion Criteria:

* Patients with cardiogenic (acute pericarditis, rheumatic coronary arteritis, hypertrophic cardiomyopathy, etc.) Or non-cardiogenic chest pain.
* any subject who suffer from malignant tumors, infectious diseases, advanced liver disease, major disability and cannot participate in the study.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiovascular disease patients (30-85 years old) who have been living in Guangdong province for more than 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | 4 years
  All-cause mortality was confrmed through a combination of hospital medical records, telephone contacts with patients or family members, and death registration at the Guangdong Provincial Center for Disease Control and Prevention.

SECONDARY OUTCOMES:
Cardiovascular Mortality | 4 years
  Cardiovascular mortality was defned as death attributable to an ischemic cardiovascular cause (including fatal MI, stroke, and peripheral arterial disease) or sudden death due to an unknown but presumed cardiovascular cause in high-risk patients.

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, Principal Investigator — School of Public Health,Nutrition and Food Hygiene,Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Lin Y, Wang S, Zhou S, Ju J, Wang X, Chen Y, Xia M. Extracellular Superoxide Dismutase Is Associated With Left Ventricular Geometry and Heart Failure in Patients With Cardiovascular Disease. J Am Heart Assoc. 2020 Aug 4;9(15):e016862. doi: 10.1161/JAHA.120.016862. Epub 2020 Jul 29. PMID 32750295